CLINICAL TRIAL: NCT02055586
Title: A Pilot Study of FLT-PET/MRI for Early Response Monitoring to Novel Cancer Therapeutic Agents
Brief Title: FLT-PET/MRI for Early Response Monitoring to Novel Cancer Therapeutic Agents
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: CASE3Y12; NCI-2013-01177 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-02-03; First posted 2014-02-05 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — alovudine; Positron-Emission Tomography; Tomography, Emission-Computed; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Diagnostic (FLT-PET/MRI): Patients undergo FLT-PET/MRI twice at baseline and once within 4 weeks after start of treatment.
  Interventions: Other: fluorine F 18 fluorothymidine; Device: positron emission tomography; Device: magnetic resonance imaging

INTERVENTIONS:
Other: fluorine F 18 fluorothymidine — Undergo FLT-PET/MRI
  Other Names: 18F-FLT; 3'-deoxy-3'-[18F]fluorothymidine; fluorothymidine F-18
Device: positron emission tomography — Undergo FLT-PET/MRI
  Other Names: PET/MR; PET; PET scan; tomography, emission computed
Device: magnetic resonance imaging — Undergo FLT-PET/MRI
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging

SUMMARY:
This pilot clinical trial studies fluorine F 18 fluorothymidine (FLT)-positron emission tomography/magnetic resonance imaging (PET/MRI) in measuring early response in patients with metastatic solid tumors receiving treatment that blocks blood flow to the tumor. Diagnostic procedures, such as FLT-PET/MRI, may help measure a patient's response earlier during treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

The primary objective of this pilot imaging study is to determine the feasibility of FLTPET/MR imaging for early prediction of treatment response in patients undergoing antiangiogenic cancer treatment. The study will assess PET/MRI test-retest reproducibility and compare baseline PET/MRI with PET/MRI after initiation (within 2-4 weeks) of antiangiogenic therapy.

SECONDARY OBJECTIVES:

* To compare early changes in PET biomarker (FLT) tumor uptake with treatment response assessed at completion of therapy (prediction of treatment response).
* To compare changes in MRI signal intensities (multi-parametric MRI) with treatment response assessed at completion of therapy.
* To compare results from multi-parametric MR imaging with FLT tumor uptake.
* To assess combinations of quantitative PET and MRI metrics.

OUTLINE:

Patients undergo FLT-PET/MRI twice at baseline and once within 4 weeks after start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic solid tumors scheduled to undergo treatment with novel cancer therapeutic agents as standard of care (SOC) treatment.
* Patients able to tolerate PET/MRI scans
* Informed consent must be given and signed

Exclusion Criteria:

* Subjects who do not meet the above mentioned inclusion criteria
* Subjects who refuse to give and/or sign the informed consent
* Patients who currently have a pacemaker
* Patients who have a history of serious adverse events related to a previous MRI or PET/CT
* Patients who are unable to undergo MRI scanning due to exclusion by UHCMC MRI restriction policies as mentioned in the standard UHCMC MRI informed consent form
* Patients with a known allergy against any component of the contrast enhancing agent
* Patients who currently pregnant or breast feeding; negative serum pregnancy test within 72 hours of their first FLT-PET/MRI
* Anti-cancer treatment (chemotherapy and/or radiation therapy) within the last 4 weeks
* Renal insufficiency: elevated creatinine and/or glomerular filtration rate (GFR) < 40 ml/min/1.73^2 (exclusion criterion only for contrast enhanced MRI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic solid tumors scheduled to undergo treatment with novel cancer therapeutic agents as SOC treatment at a cancer center hospital
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-10-22 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2017-12-27 (Actual)

PRIMARY OUTCOMES:
Concordance analysis of standardized uptake values (SUVs) between the 2 baseline scans | Baseline
  A sample size of 20 produces a two-sided 95% confidence interval [0.553, 0.918] for the Pearson correlation coefficient when the sample correlation is 0.80. Additional analysis for concordance will include Bland-Altman plots and intraclass correlation.
Comparative Analysis of PET/MRI Images | Up to 4 weeks
  Describe changes in images at baseline PET/MRI scan compared to PET/MRI image taken after initiation of anti-angiogenic therapy

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Avril, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Comprehensive Cancer Center, Cleveland, Ohio, United States